CLINICAL TRIAL: NCT00509977
Title: A Randomized, Rater-blinded, Split-face Comparison of the Efficacy of Intense Pulse Light vs. Q-switched Nd:Yag Laser for the Treatment of Melasma.
Brief Title: Study of Light Treatment and Laser Treatment for Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU706
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Light therapy
  Interventions: Procedure: Light Treatment
- 2 (Experimental): Laser Treatment
  Interventions: Procedure: Laser Treatment

INTERVENTIONS:
Procedure: Light Treatment — Light treatment applied to half of the face at each study visit
  Arms: 1
Procedure: Laser Treatment — Laser treatment applied to half of the face at each study visit
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy of light treatment and laser treatment for melasma. These treatment options have not been thoroughly explored in the treatment of melasma. By studying the effect of different treatments, a better treatment plan may be developed for people with melasma.

DETAILED DESCRIPTION:
The objective of this study is to determine the efficacy of light treatment and laser treatment for melasma. These treatment options have not been thoroughly explored in the treatment of melasma. By studying the effect of different treatments, a better treatment plan may be developed for people with melasma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melasma lesion measuring at least 4 square centimeters.
* Age 18-75 years.
* Good health.
* Willingness and ability to understand and provide informed consent for participation in the study.
* Ability to communicate with the investigator.
* Must be willing to forgo other treatment options for melasma during the course of the study.

Exclusion Criteria:

* Inability to understand the protocol or to give informed consent.
* Mental illness.
* Under 18 years of age and over 75 years of age.
* Laser treatment in the last 6 months before enrollment.
* Isotretinoin within the past year.
* Lidocaine allergy.
* History of herpes simplex viral infection.
* Concurrent active disease to facial area (i.e acne).
* Bleeding disorder.
* History of abnormal wound healing.
* History of abnormal scarring.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Melasma Area and Severity Index | 20 weeks

SECONDARY OUTCOMES:
Safety | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Collyer J, Boone SL, White LE, Rademaker A, West DP, Anderson K, Kim NA, Smith S, Yoo S, Alam M. Comparison of treatment of cherry angiomata with pulsed-dye laser, potassium titanyl phosphate laser, and electrodesiccation: a randomized controlled trial. Arch Dermatol. 2010 Jan;146(1):33-7. doi: 10.1001/archdermatol.2009.318. PMID 20083690